CLINICAL TRIAL: NCT00446498
Title: Continuous Positive Airway Pressure Versus Non-Invasive Positive Pressure Support Ventilation in Acute Cardiogenic Pulmonary Oedema: a Prospective Randomised Multicentre Trial.
Brief Title: CPAP Versus NPPV in ACPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale S. Giovanni Bosco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gbosco1
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2007-04-03 (Estimated); Status verified 2007-04

CONDITIONS: Pulmonary Edema
MeSH Terms: conditions — Pulmonary Edema | interventions — Continuous Positive Airway Pressure; Noninvasive Ventilation

INTERVENTIONS:
Device: CPAP and Non Invasive Ventilation

SUMMARY:
To assess the intubation rate in patients affected by severe cardiogenic pulmonary edema treated with CPAP or NPPV.

DETAILED DESCRIPTION:
Background Although non-invasive ventilation has shown to be an effective treatment for acute cardiogenic pulmonary oedema (ACPO), literature still lacks of multi-centre randomised prospective studies that compares CPAP with NPPV.

Aim of the study was to assess efficacy and safety of CPAP and NPPV in patients with ACPO.

Methods 80 patients with ACPO were randomly assigned to receive CPAP or NPPV (40 for each group) through a face mask.

Inclusion criteria were: severe dyspnoea, respiratory rate > 30, PaO2/FiO2 < 200, muscle fatigue.

Main end-points were endotracheal intubation, length of ventilation, hospital length of stay and mortality.

ELIGIBILITY:
Inclusion Criteria:

* rapid onset of the symptoms
* severe dyspnoea at rest
* respiratory rate > 30 breath per minute
* use of accessory respiratory muscles
* PaO2/FiO2 < 200, radiological findings of ACPE

Exclusion Criteria:

* ST elevation myocardial infarction
* hemodynamic instability (systolic arterial pressure < 90 mmHg
* need for immediate endotracheal intubation (respiratory arrest, bradypnea
* inability to protect the airways, impaired sensorium (agitation or unconsciousness
* inability to clear secretions, respiratory tract infections
* chronic obstructive pulmonary disease (COPD) exacerbation, chronic respiratory failure necessitating long-term oxygen therapy
* pulmonary embolism, pneumonia, recent oesophageal-gastric surgery
* gastrointestinal bleeding
* facial deformities
* haematological malignancy or cancer with Eastern Cooperative Oncology Group (ECOG) performance status ≥ 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2002-07; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Intubation rate

SECONDARY OUTCOMES:
time of recovery
hospital length of stay
mortality and improvement in gas exchange

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Ferrari, MD, Principal Investigator — Ospedale San Giovanni Bosco ASL4; Giovanni Ferrari, MD, Principal Investigator — Ospedale San Giovanni Bosco ASL4 Torino Italy
Locations (1):
- Ospedale San Giovanni Bosco Medicina d'Urgenza, Torino, Italy